CLINICAL TRIAL: NCT02173457
Title: Phase III Study of Chiglitazar in Patients With Type 2 Diabetes Mellitus and Insufficient Glycemic Control Despite Diet and Exercise -- A Multicenter, Randomized, Double-Blind, and Sitagliptin-Controlled Trial
Brief Title: Study of Chiglitazar Compare With Sitagliptin in Type 2 Diabetes Patients
Acronym: CMAS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chipscreen Biosciences, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CGZ302
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
Keywords: Chiglitazar; Sitagliptin; diabetes; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — chiglitazar; Sitagliptin Phosphate; 4-Acetamido-4'-isothiocyanatostilbene-2,2'-disulfonic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Patients administrate Chiglitazar 32mg once daily for 24 weeks
  Interventions: Drug: Chiglitazar
- Arm 2 (Experimental): Patients administrate Chiglitazar 48mg once daily for 24 weeks
  Interventions: Drug: Chiglitazar
- Arm 3 (Active Comparator): Patients administrate Sitagliptin 100mg once daily for 24 weeks
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Chiglitazar — Take orally
  Other Names: CS038
  Arms: Arm 1; Arm 2
Drug: Sitagliptin — Take orally
  Other Names: Sit
  Arms: Arm 3

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Chiglitazar, compare with Sitagliptin.

DETAILED DESCRIPTION:
The efficacy and safety will be compared between Chiglitazar and Sitagliptin after treatment of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the WHO Diagnostic Criteria for Type 2 Diabetes (published on 1999);
2. HbA1c≥ 7.5% and ≤ 10.0% after control of diet and exercises;
3. Male and female,age between 18 and 70 years;
4. BMI between 18.5-35kg/m2;
5. Willing to be assigned to any treatment arm and sign inform consent.

Exclusion Criteria:

1. Type 1 diabetes;
2. Treated by oral or injective antidiabetic drug before screening, including insulin and herb;
3. Fasting plasma glucose > 13.3 mmol/L (240 mg/dL);
4. Resistant hypertension [blood pressure above the goal despite adherence to at least 3 optimally dosed antihypertensive medications (including diuretic) of different classes,or blood pressure is controlled to below the goal by at least different classes of drugs];
5. Plasma triglyceride > 500 mg/dL (5.65 mmol/L);
6. Is treating by fibrates;
7. History of diabetic ketoacidosis,diabetic hyperglycemic hyperosmolar syndrome,lactic acidosis, diabetic hypoglycemia; or is currently combined with retinopathy, diabetic nephropathy and diabetic neuropathy;
8. Had transient ischemic attack,cerebrovascular accident or unstable angina in the past 6 months;
9. History of myocardial infarction or had conducted coronary angioplasty or coronary artery bypass graft surgery;
10. Had or is having pancreatic diseases;
11. Heart failure (NYHA classification Stage III or IV), or left ventricular hypertrophy indicated by ECG;
12. Hepatic diseases such as hepatocirrhosis, active hepatitis,aspartate aminotransferase or alanine aminotransferase > 2.5 fold of the upper limit of the normal range;
13. Kidney diseases or serum creatinine exceed the normal range: male > 133 μmol/L or female >108 μmol/L;
14. Had malignancy in the past 5 years, not including basal cell carcinoma;
15. Had or is currently receiving treatment that can alter blood glucose metabolism, including but not limited to diuretic,hormone (corticotropin or steroids),beta blockers;
16. Have the diseases that can alter blood glucose metabolism, including but not limited to active hepatitis, hyperthyroidism,or adrenal tumors;
17. Edema with unknown reason;
18. Alcohol or drug addiction;
19. Had participated other drugs' clinical trials in the 3 months before screening;
20. Pregnant or lactic women; or women of childbearing age who are not able to or is not willing to conduct contraception;
21. Any condition that make investigator consider the subject is not suitable to participate the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline after 24 weeks of treatment | 24 weeks
  The change of HbA1c at week 24 from baseline

SECONDARY OUTCOMES:
Change in HbA1c from baseline for patients with a baseline HbA1c >=8.5% | 24 weeks
  The change of HbA1c at week 24 from baseline for patients with a HbA1c >=8.5% at baseline
Change in HbA1c from baseline for patients with a baseline HbA1c <8.5% | 24 weeks
  The change of HbA1c at week 24 from baseline for patients with a HbA1c < 8.5% at baseline
Change in HbA1c from baseline | 12 weeks
  The change of HbA1c at week 12 from baseline
Percentage of patients that attained target HbA1c <7.0% | 24 weeks
  Percentage of patients whose HbA1c at week 24 are < 7.0%
Percentage of patients whose HbA1c lowered by at least 0.5% | 24 weeks
  Percentage of patients whose change of HbA1c at week 24d from baseline are >= 0.5%
Change in fasting plasma glucose from baseline | 12 and 24 weeks
  The change of fasting plasma glucose at week 12 and 24 from baseline
Change in 2-h postprandial glucose (2hPPG) from baseline | 12 and 24 weeks
  The change of 2-h postprandial glucose (2hPPG) at week 12 and 24 from baseline
Change in total cholesterol (TC) from baseline | 12 and 24 weeks
  The change of total cholesterol (TC) at week 12 and 24 from baseline
Change in triglyceride from baseline | 12 and 24 weeks
  The change of triglyceride at week 12 and 24 from baseline
Change in high density lipoprotein cholesterol (HDL-C) from baseline | 12 and 24 weeks
  The change of high density lipoprotein cholesterol (HDL-C) at week 12 and 24 from baseline
Change in low density proprotein cholesterol (LDL-C) from baseline | 12 and 24 weeks
  The change of low density lipoprotein cholesterol (LDL-C) at week 12 and 24 from baseline
Change in free fatty acid (FFA) from baseline | 12 and 24 weeks
  The change of free fatty acid (FFA) at week 12 and 24 from baseline
Change in fasting plasma insulin from baseline | 12 and 24 weeks
  The change of fasting plasma insulin at week 12 and 24 from baseline
Insulin sensitivity assessed by the homeostatic model assessment (HOMA) at 12 and 24 weeks, compared with that of baseline | 12 and 24 weeks
  The change of insulin sensitivity at week 12 and 24 from baseline
Change in blood pressure from baseline | 24 weeks
  The change of blood pressure at week 24 from baseline
Percentage of patients who discontinue the trial due to hyperglycemia | 24 weeks
  The percentage of patients who discontinue the trial due to hyperglycemia during the 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, Dr., Principal Investigator — Shanghai 6th People's Hospital
Locations (37):
- China (37):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Hospital Affiliated to Anhui Medical University, Hefei, Anhui
  - Fuwai Hospital, Beijing, Beijing Municipality
  - The General Hospital of the Chinese People's Armed Police Forces, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - The Second Artillery General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Affiliated to Capital Medical Universtiy, Beijing, Beijing Municipality
  - The Third Hospital Affiliated to Guangzhou Medical College, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Beijing University Shenzhen Hospital, Shenzhen, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University (The Eastern Hospital), Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University (The Western Hospital), Nanning, Guangxi
  - The Second Hospital of Heibei Medical University, Shijiazhuang, Hebei
  - Tongji Hospital Affiliated to Tongji Medical College of HUST, Wuhan, Hubei
  - The First Hospital Affiliated to Nanhua University, Hengyang, Hunan
  - The First People's Hospital of Yueyang, Yueyang, Hunan
  - The Affiliated Hospital of Inner Mongolia, Hohhot, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Gulou Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - The Second Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shan'xi
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - The Qingpu Branch of Zhongshan Hospital Affiliate to Fudan University, Shanghai, Shanghai Municipality
  - Tongji Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai 5th People's Hospital, Shanghai, Shanghai Municipality
  - The Central Hospital of Minhang District of Shanghai, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Zhou Y, Zhou X, Su X, Xu X, Li H, Ma J. Effect of Chiglitazar and Sitagliptin on Bone Mineral Density and Body Composition in Untreated Patients with Type 2 Diabetes. Diabetes Metab Syndr Obes. 2023 Dec 27;16:4205-4214. doi: 10.2147/DMSO.S439479. eCollection 2023. PMID 38162801
- [Derived] Zhou Y, Wang H, Wang Y, Xu X, Li F, Zhou J, Shan T, Huang R, Cai T, Liu X, Su X, Li H, Ma J. Comparative Evaluation of Chiglitazar and Sitagliptin on the Levels of Retinol-Binding Protein 4 and Its Correlation With Insulin Resistance in Patients With Type 2 Diabetes. Front Endocrinol (Lausanne). 2022 Apr 25;13:801271. doi: 10.3389/fendo.2022.801271. eCollection 2022. PMID 35547000